CLINICAL TRIAL: NCT03169582
Title: Avanafil Versus Sildenafil in Spinal Cord Injury Erectile Dysfunction: Non- Inferiority, Randomized, Crossover, Open Clinical Trial
Brief Title: Avanafil Versus Sildenafil in Spinal Cord Injury Erectile Dysfunction
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Eduardo Vargas-Baquero (Other)
Responsible Party: Sponsor-Investigator, Eduardo Vargas-Baquero, Principal Investigator, Hospital Nacional de Parapléjicos de Toledo
Organization: Hospital Nacional de Parapléjicos de Toledo (Other)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: HNParaplejicos
Record Dates: First submitted 2017-04-21; First posted 2017-05-30 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — avanafil; Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: non- inferiority, randomized, crossover, open clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Avanafil (Active Comparator): Clinical evaluation of the two pharmacological interventions (Sildenafil vs Avanafil).
  Interventions: Drug: Avanafil
- Sildenafil (Active Comparator): Clinical evaluation of the two pharmacological interventions (Sildenafil vs Avanafil)
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Avanafil — Drug administration (Avanafil)
  Other Names: no other interventions
  Arms: Avanafil
Drug: Sildenafil — Drug administration (Sildenafil)
  Other Names: no other interventions
  Arms: Sildenafil

SUMMARY:
The main goal of this study is to compare the use of Avanafil versus Sildenafil in spinal cord injury erectile dysfunction. The study has the characteristics of a non- inferiority, randomized, crossover, open clinical trial. The principal variable is the IIEF-EF (Erectile Function Domain questionnaire of the International Index of Erectile Function IIEF).

This is an interventional study

ELIGIBILITY:
Inclusion Criteria:

* Spinal cord injury
* Erectile dysfunction
* No Medical Contraindication to use Avanafil and/or Sildenafil
* Able to provide informed consent
* Able to complete questionnaires

Exclusion Criteria:

* Medical Contraindication to use Avanafil and/or Sildenafil
* No spinal cord injury
* Congenital spinal cord injury
* Not able to provide informed consent
* Not able to complete questionnaires

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Estimated)
Dates: Start 2016-04-01 (Actual); Primary Completion 2018-06-01 (Estimated); Study Completion 2018-06-01 (Estimated)

PRIMARY OUTCOMES:
IIEF-EF | 2 years
  Erectile Function Domain questionnaire of the International Index of Erectile Function.

SECONDARY OUTCOMES:
SLQQ-Part II | 2 years
  Sexual life quality Questionnaire
GAQ | 2 years
  Global Impression of efficacy

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Nacional de Paraplejicos, Toledo, Spain

IPD SHARING:
Plan to Share IPD: No